CLINICAL TRIAL: NCT06639698
Title: Treatment of Menstrual Cycle Alterations in Women With PCOS of Phenotype D Using Dietary Supplementation That Combines Diosgenin, Vitamin D and Alpha-lactalbumin
Brief Title: Treatment of Women With PCOS of Phenotype D
Acronym: PT-PHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILOT-PHD-129
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: PCOS phenotype D; Diosgenin; Dioscorea
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diosgenin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients will take a tablet containing diosgenin (120 mg), alpha-lactalbumin (100 mg) and vitamin D (50 mcg) - two times per day for six months
  Interventions: Dietary Supplement: Diosgenin

INTERVENTIONS:
Dietary Supplement: Diosgenin — Patients will take a tablet containing diosgenin (120 mg), alpha-lactalbumin (100 mg) and vitamin D (50 mcg) - two times per day for six months

SUMMARY:
In this study, female patients diagnosed with PCOS of phenotype D will be enrolled. They generally display the following characteristics: menstrual cycle alterations; polycystic ovary morphology at ultrasound; normal blood levels of androgen, particularly testosterone; no signs of clinical hyperandrogenism.

Current treatments for this condition include insulin sensitizers (such as metformin) and hormonal contraceptives. However, this specific phenotype of PCOS do not feature metabolic or hormonal alterations, and the efficacy of these treatments has lately been questioned.

In the present clinical trial, patients will be given a dietary supplement containing Dioscorea extract (source of Diosgenin, a natural analog of progesterone), vitamin D and alpha-lactalbumin for six month. Restoration of regular menstrual cycle and physiological ultrasound appearance of the ovaries will be the primary goal of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS of phenotype D, according to the Rotterdam Criteria and the EGOI-PCOS Criteria

Exclusion Criteria:

* Diagnosis of PCOS of phenotype A, B or C, according to the Rotterdam Criteria and the EGOI-PCOS Criteria
* Hormonal treatments;
* Treatments with inositol or other insulin sensitizers (such as metformin);
* Insulin resistance or pre-diabetes condition
* BMI > 30
* Endocrinological alterations
* Chronic pharmacological therapies
* Major pathological conditions (e.g. tumors or autoimmune diseases)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Restoration of regular menstrual cycle | From enrollment (T0) to the completion of the study at 6 months (T6M)
  Restoration of regular menstrual cycle will be assessed counting the days between two subsequent menstrual cycles, using a menstrual diary updated by the patients

SECONDARY OUTCOMES:
Restoration of physiological appearance of the ovaries at ultrasound | From enrollment (T0) to the completion of the study at 6 months (T6M)
  Reduction of the ultrasonography count of arrested ovarian follicles

CONTACTS AND LOCATIONS:
Locations (1):
- Alma Res Fertility Center, Rome, ITA, Italy